CLINICAL TRIAL: NCT06943157
Title: Investigation of the Relationship Between Self-Efficacy and Adherence to Medication in Individuals With Coronary Artery Disease: A Descriptive and Correlational Study
Brief Title: Self-Efficacy and Medication Adherence in Patients With Coronary Artery Disease: A Descriptive Study
Acronym: SEMACAD
Status: Recruiting | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Zeynal KİZİR, PhD Student, Hasan Kalyoncu University, Faculty of Health Sciences, Nursing Department, Hasan Kalyoncu University
Other Study IDs: HKU-KAH-2025-01
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease
Keywords: Nurse; Coronary Artery Disease; Self-Efficacy; Medication Adherence
MeSH Terms: conditions — Coronary Artery Disease; Medication Adherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease Patients: This cohort consists of individuals aged 18 and older who have been diagnosed with coronary artery disease for at least one year and are being followed in cardiology or cardiovascular surgery outpatient or inpatient clinics. Patients included are those who volunteered to participate in the study, can communicate in Turkish, and do not have any mental disorders.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a descriptive, observational study. No intervention or experimental procedure was performed. Data were collected using self-administered questionnaires without influencing participant behavior or treatment.

SUMMARY:
This descriptive study aims to examine the relationship between self-efficacy and medication adherence in individuals with coronary artery disease (CAD). The study will be conducted between March and October 2025 at Adıyaman University Training and Research Hospital with a planned sample size of 135 participants. Data will be collected using a Descriptive Information Form, the Self-Efficacy for Managing Chronic Disease Scale, and the Medication Adherence Report Scale (MARS).

DETAILED DESCRIPTION:
Coronary artery disease (CAD) remains one of the leading causes of death worldwide. Managing CAD requires long-term treatment adherence and lifestyle changes. Self-efficacy, which reflects an individual's belief in their ability to perform specific health behaviors, plays a key role in disease management. In CAD patients, high levels of self-efficacy have been associated with better treatment adherence, improved symptom management, and successful adoption of healthy behaviors.

This descriptive study is designed to investigate the relationship between self-efficacy and medication adherence in individuals diagnosed with CAD. The study will be carried out at Adıyaman University Training and Research Hospital between March and October 2025. The target population includes patients who have been diagnosed with CAD (e.g., angina pectoris, myocardial infarction) for at least one year and meet the inclusion criteria. Based on a power analysis using G*Power software (effect size f² = 0.15, α = 0.05, power = 0.90), the required sample size is calculated as 112. However, accounting for possible data loss or participant dropout, the final sample size is set at 135.

Data collection tools include:

Descriptive Information Form to assess demographic and clinical characteristics,

The 6-Item Self-Efficacy for Managing Chronic Disease Scale, validated in Turkish by İncirkuş and Özkan Nahcivan (Cronbach's alpha = 0.90),

Medication Adherence Report Scale (MARS), adapted to Turkish by Temeloğlu Şen et al. (Cronbach's alpha = 0.78).

The findings are expected to contribute to the literature and guide healthcare professionals, particularly nurses, in planning educational and counseling services to improve self-efficacy and medication adherence among CAD patients.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older

Having been diagnosed with Coronary Artery Disease (angina pectoris, unstable angina, myocardial infarction) at least 1 year ago

Being followed

Being able to communicate in Turkish

Voluntarily agreeing to participate in the study

Having no diagnosed mental disorder

Exclusion Criteria:

* Having a primary diagnosis other than Coronary Artery Disease

Being unable to complete the questionnaires due to mental health problems

Providing incomplete data or withdrawing from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals aged 18 and older who have been diagnosed with coronary artery disease for at least one year and are being followed in cardiology or cardiovascular surgery outpatient/inpatient clinics at Adıyaman University Training and Research Hospital. All participants must be able to communicate in Turkish, have no diagnosed mental disorder, and voluntarily agree to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy score for chronic disease management | At the time of data collection (March 2025 - October 2025)
  Self-efficacy levels of patients with coronary artery disease will be measured using the 6-Item Self-Efficacy Scale for Chronic Disease Management. Each item is rated from 1 to 10. The total score ranges from 6 to 60, and higher scores indicate better self-efficacy in chronic disease management.

SECONDARY OUTCOMES:
Medication adherence score | At the time of data collection (March 2025 - October 2025)
  Patients' adherence to their prescribed medication regimen will be assessed using the Medication Adherence Report Scale (MARS). The MARS scale ranges from 5 to 25, with higher scores indicating better medication adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Adiyaman University Training and Research Hospital, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data (IPD).

REFERENCES:
- [Background] Fors A, Ulin K, Cliffordson C, Ekman I, Brink E. The Cardiac Self-Efficacy Scale, a useful tool with potential to evaluate person-centred care. Eur J Cardiovasc Nurs. 2015 Dec;14(6):536-43. doi: 10.1177/1474515114548622. Epub 2014 Aug 22. PMID 25149667